CLINICAL TRIAL: NCT00442962
Title: The Effect of Prior Short Course Combination Antiretroviral Therapy Administered for the Prevention of Mother-to-Child Transmission (pMTCT) of HIV-1 on Subsequent Treatment Efficacy in Treatment-"Nearly Naive" Participants
Brief Title: HIV Treatment Reinitiation in Women Who Received Anti-HIV Drugs to Prevent Mother-to-Child Transmission of HIV
Acronym: Nearly Naive
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5227; 1U01AI068636 (NIH)
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EFV + FTC/TDF (Experimental): Participants will efavirenz (600mg in pill form, taken orally, once daily) and emtricitabine/tenofovir disoproxil fumarate (200/300mg in pill form, taken orally, once daily), for 48 weeks
  Interventions: Drug: Efavirenz; Drug: Emtricitabine/Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Efavirenz — 600-mg tablet taken orally daily
  Other Names: EFV
Drug: Emtricitabine/Tenofovir disoproxil fumarate — 200-mg emtricitabine/300-mg tenofovir disoproxil fumarate tablet taken orally once daily
  Other Names: Truvada

SUMMARY:
The purpose of this study is to determine if pregnancy-limited, short-term combination HIV treatment regimens -- which were used solely for the prevention of mother to child transmission of HIV and discontinued postpartum -- decreases the effectiveness of a standard initial regimen of anti-HIV drugs when subsequent treatment is needed.

DETAILED DESCRIPTION:
Stopping and restarting highly active antiretroviral therapy (HAART) is not generally recommended because it has the potential to allow drug-resistant HIV to emerge. However, to prevent mother-to-child transmission (MTCT), HIV infected women who are pregnant are temporarily put on HAART, even if HIV treatment is not indicated at the time. It is unknown if such short-term therapy affects the viral response to HAART later, when permanent therapy is clinically indicated. The purpose of this study is to determine if HAART taken to prevent MTCT during pregnancy has an effect on the ability of a standard initial regimen of HAART to suppress HIV viral load.> >>

>

>> Study follow-up will last for 48 weeks per participant. Participants will take a daily regimen of efavirenz and emtricitabine/tenofovir disoproxil fumarate. There will be 8 clinical visits in this study; visits will occur at baseline and at Weeks 2, 4, 8, 16, 24, 36, and 48. At each visit, a physical exam, blood and urine collection, and pregnancy tests will occur. At some visits, adherence, quality-of-life, and birth control interviews will be completed.>

>>

>

>> Enrollment in this study will last until 47 participants have joined or until December 31, 2009, whichever comes later.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Viral load of 500 copies/mL or more
* Prior HAART for more than 7 days, but less than 40 weeks during at least one previous pregnancy for prevention of MTCT of HIV
* Clinical or laboratory indication to start HAART, in the opinion of the participant's physician
* Certain laboratory values
* Willingness to use acceptable forms of contraception
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Taking any antiretroviral medication within 24 weeks prior to study entry
* Evidence of certain HIV-1 RT mutations within 90 days prior to study entry (version 1.0)
* Evidence of certain HIV-1 RT mutations identified by standard bulk viral population genotypic resistance tests at any time prior to study entry, if available (version 2.0, 09/03/2009)
* Treatment at any time, for any reason with nevirapine as a single agent OR addition of any part of the study regimen as a single agent to a failing regimen
* Use of certain antihistamines, certain anti-infectives, cisapride, St John's wort, midazolam, triazolam, dihydroergotamine, ergonovine, ergotamine, or methylergonovine within 14 days prior to study entry
* Use of HIV vaccine, chronic systemic corticosteroids, interleukins, interferons, other cytokines, or investigational therapy within 30 days prior to study entry
* Acute or chronic therapy for certain serious medical illnesses within 14 days of study entry. Participants who have completed 7 days of therapy and are judged clinically stable are not excluded.
* Cancer requiring systemic chemotherapy
* Known allergy/sensitivity to the study drugs or their formulations
* Current drug or alcohol use that, in the opinion of the investigator, would interfere with the study
* Two consecutive HIV viral loads of more than 5,000 copies/mL 8 weeks or more following initiation of HAART during pregnancy and while still receiving HAART
* Two consecutive viral loads of more than 400 copies/mL 24 weeks or more following initiation of HAART during pregnancy while still receiving HAART
* Current imprisonment or involuntary incarceration in a medical facility for psychiatric or physical illness
* Pregnancy or breastfeeding

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary A. Vogler, MD, Study Chair — Division of Infectious Diseases, Weill College of Medicine of Cornell University
Locations (9):
- United States (6):
  - Ucsd, Avrc, San Diego, California
  - Brigham and Women's Hospital, Division of Infectious Disease, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Med. College of Cornell Univ., The Cornell CTU -Chelsea, New York, New York
  - Bronx-Lebanon Hosp. Ctr. CRS, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
- Instituto de Pesquisa Clinica Evandro Chagas Fiocruz, Fundacao Oswaldo Cruz, Rio de Janeiro, Brazil
- Peru (2):
  - San Miguel CRS, San Miguel, Lima region
  - Barranco CRS, Lima

REFERENCES:
- [Background] Abrams EJ. Prevention of mother-to-child transmission of HIV--successes, controversies and critical questions. AIDS Rev. 2004 Jul-Sep;6(3):131-43. PMID 15595430
- [Background] Bassetti D, Cargnel A. Genotypic resistance tests for the management of the HIV-infected pregnant woman. Scand J Infect Dis Suppl. 2003;106:70-4. PMID 15000589
- [Background] Duran AS, Losso MH, Salomon H, Harris DR, Pampuro S, Soto-Ramirez LE, Duarte G, de Souza RS, Read JS; NISDI Perinatal Study Group. Drug resistance among HIV-infected pregnant women receiving antiretrovirals for prophylaxis. AIDS. 2007 Jan 11;21(2):199-205. doi: 10.1097/QAD.0b013e328011770b. PMID 17197811
- See also: Click here for more information on this network of studies — http://www.actgnetwork.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at 8 sites from 3 countries: 6 in the US, 1 in Brazil, 1 in Peru, between May 2007 to December 2009.
Pre-assignment Details: HIV-infected women, at least 16 years of age, whose only prior exposure to anti-retrovirals (ARVs) was for the purpose of prevention of mother-to-child transmission, who now qualify to start ARVs for their own health.
Groups:
- EFV + FTC/TDF: Participants will take a daily regimen of efavirenz and emtricitabine/tenofovir disoproxil fumarate for 48 weeks
Period: Overall Study
Arm/Group | EFV + FTC/TDF
Started | 54
Primary Outcome Evaluation | 52 (Primary outcome evaluation at week 24.)
Completed | 46 (Completed 48 weeks of follow-up.)
Not Completed | 8
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (7)
Age, Customized [Number; unit: participants]
  Between 19 and 25 years | 19
  Between 26 and 30 years | 16
  Between 31 and 35 years | 9
  Between 36 and 40 years | 6
  Between 40 and 45 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
  Brazil | 22
  Peru | 20
CD4 count, Continuous [Mean (Standard Deviation); unit: cells/mm^3] | 264 (104)
CD4 count, Categorical [Number; unit: participants]
  < 50 cells/mm^3 | 1
  Between 50 and 99 cells/mm^3 | 0
  Between 100 and 199 cells/mm^3 | 15
  Between 200 and 299 cells/mm^3 | 18
  Between 300 and 399 cells/mm^3 | 15
  400 or more cells/mm^3 | 5
Plasma HIV-1 RNA, Continuous [Mean (Standard Deviation); unit: log10 copies/mL] | 4.5 (0.6)
Plasma HIV-1 RNA, Categorical [Number; unit: participants]
  <= 400 copies/mL | 0
  Between 401 and 1000 copies/mL | 1
  Between 1001 and 10,000 copies/mL | 8
  Between 10,001 and 50,000 copies/mL | 20
  Between 50,001 and 75,000 copies/mL | 11
  Between 75,001 and 250,000 copies/mL | 12
  More than 250,000 copies/mL | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Early Virologic Response
Description: Plasma HIV-1 Viral Load Fewer Than 400 Copies/ml
Time Frame: At Week 24
Population: Intention to treat (ignoring current study treatment status or history); closest measurement to week 24 used; missing measurements ignored. Exact binomial confidence interval calculated using method of Blyth-Still-Casella.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 52
percentage of participants | 80.8 [67.8 to 90.4]

2. Secondary Outcome: Time to First Safety Event
Description: Time from starting study treatment to first grade 3 or 4 sign/symptom or laboratory abnormality and at least one grade higher than baseline. Grading used the Division of AIDS (DAIDS) 2004 Severity of Adverse Events Tables.
Time Frame: Throughout study
Population: All enrolled participants who started study treatment (which in this case, matches the number of participants enrolled.)
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 54
weeks
  5th percentile | 4.1 [0.9 to 24.4]
  10th percentile | 24.4 [0.9 to NA] — Not estimable as the upper limit for survival function at all weeks is above 90%
  15th percentile | 33.1 [4.1 to NA] — Not estimable as the upper limit for survival function at all weeks is above 85%

3. Secondary Outcome: Percentage of Participants With Early Virologic Suppression
Description: Plasma HIV-1 Viral Load Fewer Than 50 Copies/ml
Time Frame: At Weeks 24
Population: ITT (ignoring current study treatment status and history); missing values ignored and closest value to week 24 used if multiple results available. 2 fewer results available compared to primary outcome b/c testing by ultrasensitive assay may have been retrospective.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 50
percentage of participants | 72.0 [58.7 to 83.8]

4. Secondary Outcome: Percentage of Participants With Late Virologic Response
Description: Plasma HIV-1 Viral Load Fewer Than 400 Copies/ml
Time Frame: At Week 48
Population: Participants with plasma HIV-1 RNA viral load result available from week 48 study visit.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 46
percentage | 80.43 [67.1 to 89.7]

5. Secondary Outcome: Time to Initial Virologic Response
Description: Time from enrollment to scheduled week of first plasma HIV-1 RNA viral load fewer than 400 copies/mL.
Time Frame: Throughout study
Population: All enrolled participants included.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 54
weeks
  50th percentile | 2 [2 to 4]
  75th percentile | 8 [4 to 16]
  95th percentile | 24 [16 to NA] — Not estimable as the upper limit for survival function at all weeks is above 95%

6. Secondary Outcome: Time to Initial Virological Failure
Description: Virologic failure defined as two consecutive measurements of plasma HIV-1 RNA at least 400 copies/mL at or after the week 16 study visit. Time measured from enrollment.
Time Frame: Throughout study
Population: All participants enrolled are included.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 54
weeks
  5th percentile | 16 [16 to 16]
  10th percentile | 16 [16 to 36]
  15th percentile | 24 [16 to NA] — Not estimable as the upper limit for survival function at all weeks is above 85%

7. Secondary Outcome: Time to Loss of Virologic Response by Week 48 (Defined by FDA TLOVR Algorithm)
Time Frame: Throughout study
Population: All enrolled participants included.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 54
weeks
  10th percentile | 16 [0 to 24]
  15th percentile | 24 [0 to 36]
  20th percentile | 24 [4 to NA] — Not estimable as the upper limit for survival function at all weeks is above 80%

8. Secondary Outcome: Early Changes in CD4 Count From Baseline
Description: Changes in CD4+ lymphocyte counts between study visit weeks 4, 8 16 and 24 and baseline.
Time Frame: At weeks 0(baseline), 4, 8, 16, 24
Population: Intent to treat (study treatment status and history ignored); missing measurements ignored.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 51
cells/mm^3
  Change from baseline to week 4 | 105 (108)
  Change from baseline to week 8 | 118 (87)
  Change from baseline to week 16 | 138 (112)
  Change from baseline to week 24 | 147 (147)

9. Secondary Outcome: Percentage of Participants With Late Virologic Suppression
Description: Plasma HIV-1 Viral Load Fewer Than 50 Copies/ml
Time Frame: At Week 48
Population: Participants with ultra-sensitive (detectable to 50 copies/mL) plasma HIV-1 RNA result available from week 48 visit.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 44
percentage | 70.5 [55.8 to 82.1]

10. Secondary Outcome: Time to First Dose Modification
Description: Time from starting study treatment to first dose/drug modification.
Time Frame: Throughout study
Population: All enrolled participants who started study treatment.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 54
weeks
  10th percentile | 1.9 [0.4 to 25.7]
  15th percentile | 24.9 [1.1 to 39.1]
  20th percentile | 25.7 [1.9 to NA] — Not estimable as the upper limit for survival function at all weeks is above 80%

11. Secondary Outcome: Late Change in CD4 Count From Baseline
Description: Change in CD4+ lymphocyte counts between week 48 study visit and baseline.
Time Frame: At week 48
Population: Participants with a CD4+ lymphocyte cell count result from the week 48 study visit.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | EFV + FTC/TDF
Number analyzed (Participants) | 46
cells/mm^3 | 194 (185)

ADVERSE EVENTS:
Groups:
- EFV+FTC/TDF: Participants will take a daily regimen of efavirenz and emtricitabine/tenofovir disoproxil fumarate for 48 weeks
Arm/Group | EFV+FTC/TDF
Serious Adverse Events (participants affected / at risk) | 1/54
Other Adverse Events (participants affected / at risk) | 41/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EFV+FTC/TDF (N=54)
Suicide attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EFV+FTC/TDF (N=54)
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Pyrexia (General disorders) | 5
Drug hypersensitivity (Immune system disorders) | 3
Sinusitis bacterial (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 5
Vulvovaginal candidiasis (Infections and infestations) | 6
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 4
Blood cholesterol (Investigations) | 4
Haemoglobin decreased (Investigations) | 6
Low density lipoprotein abnormal (Investigations) | 4
Neutrophil count decreased (Investigations) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 7
Somnolence (Nervous system disorders) | 5
Abnormal dreams (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 4
Dysuria (Renal and urinary disorders) | 4
Vaginal discharge (Reproductive system and breast disorders) | 6
Vulvovaginal pruritus (Reproductive system and breast disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 8
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.